CLINICAL TRIAL: NCT01012323
Title: Clinical Study to Evaluate the Efficacy, Pharmacokinetics and Safety of Immunoglobulin Intravenous (Human) 10% (NewGam) in Patients With Primary Immunodeficiency Diseases
Brief Title: A Study of NewGam, Human Immunoglobulin 10%, in Patients With Primary Immunodeficiency Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGAM-01; 2009-011434-10 (EudraCT Number)
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Primary Immunodeficiency Diseases
Keywords: PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NewGam (Experimental): Participants received NewGam 200-800 mg/kg intravenously every 3 weeks (17 infusions) or 4 weeks (13 infusions) for 1 year.
  Interventions: Biological: NewGam

INTERVENTIONS:
Biological: NewGam — The dose of NewGam, solvent/detergent treated human normal immunoglobulin 10%, remained the same throughout the study, as long as minimum trough levels of serum immunoglobulin G (IgG) was above 5 g/L. If serum IgG trough levels dropped to 5 g/L or less, the dose was to be adjusted at the investigator's discretion. NewGam was supplied as a solution for infusion.
  Other Names: Human normal immunoglobulin

SUMMARY:
The purpose of this study was to determine the efficacy of NewGam in preventing serious bacterial infections and to determine the pharmacokinetic profile of NewGam. The safety of NewGam and its effect on quality of life were also evaluated.

DETAILED DESCRIPTION:
NewGam is a new 10% human normal immunoglobulin (IVIG) solution developed by Octapharma for intravenous administration. It is supplied as a liquid formulation ready to use. The primary therapeutic use of immunoglobulins is to provide antibodies to prevent viral and bacterial diseases (replacement therapy). IVIG has proved to be useful in a variety of clinical conditions other than for replacement of immunoglobulins; IVIG exhibits an immunomodulatory effect. Children and adults with a Primary Immunodeficiency Disease (PID) have an increased risk of recurrent bacterial and viral infections that typically attack the respiratory tract (sinusitis, bronchitis, pneumonia) but can also affect the gastrointestinal tract (gastroenteritis). Theses diseases can be severe and can lead to substantial morbidity. Responses to antibacterial therapy are often poor. At present, most primary immune deficiencies are not curable, but IVIGs have been shown to decrease the total number of severe infections and the duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 2 years and ≤ 75 years.
* Confirmed diagnosis of common variable immunodeficiency (CVID) or X-linked agammaglobulinemia (XLA).
* Previously treated with a commercial immune globulin intravenous (human) every 21-28 days for at least 6 infusion intervals at a constant dose between 200 and 800 mg/kg body weight.

Exclusion Criteria:

* Acute infection requiring intravenous antibiotic treatment within 2 weeks prior to and during the screening period.
* Exposure to blood or any blood product or derivative, other than commercially available intravenous immunoglobulin (IVIG), within the past 3 months prior to enrollment.
* Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products, or any component of the investigational product.
* Requirement of any routine pre-medication for IVIG infusion.
* Severe liver function impairment (alanine aminotransferase [ALAT] 3x > upper limit of normal).
* Presence of renal function impairment (creatinine > 120 μmol/L), or predisposition for acute renal failure (eg, any degree of pre-existing renal insufficiency or routine treatment with known nephritic drugs).
* History of autoimmune hemolytic anemia.
* History of diabetes mellitus.
* Congestive heart failure New York Heart Association (NYHA) class III or IV.
* Non-controlled arterial hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 90 mmHg).
* History of deep vein thrombosis or thrombotic complications of IVIG therapy.
* A positive result at screening on any of the following viral markers: human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV).
* Treatment with steroids (oral or parenteral, long-term, ie, 30 days or more, not intermittent or burst, daily, ≥ 0.15 mg of prednisone or equivalent/kg/day), immunosuppressive or immunomodulatory drugs.
* Planned vaccination during the study period.
* Treatment with any investigational agent within 3 months prior to enrollment.
* Known or suspected to abuse alcohol, drugs, psychotropic agents or other chemicals within the past 12 months prior to enrollment.
* Pregnant or nursing women.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Sudir Gupta, MD, Irvine, California
  - Isaac Melamed, MD, Centennial, Colorado
  - James Moy, MD, Chicago, Illinois
  - William Smits, MD, Fort Wayne, Indiana
  - Dr. Alan Knutsen, St Louis, Missouri
  - Ai Lan Kobayashi, MD, Papillion, Nebraska
  - Hans Ochs, MD, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NewGam
Started | 51
Completed | 50
Not Completed | 1
Not completed — Investigator Judgment | 1

BASELINE CHARACTERISTICS:
Population: Total set: All enrolled participants.
Arm/Group | NewGam
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (19.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Bacterial Infections Per Person-year of Treatment
Description: The number of serious bacterial infections per person-year of treatment was calculated by the following formula: Total number of serious bacterial infections / patient-years on NewGam treatment. Serious bacterial infections were defined as bacteraemia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Full analysis set: All participants who received at least 1 complete treatment with NewGam and for whom data on infections were available from at least 1 post-treatment diary entry.
Measure: Number; unit: Serious infections per person-year of tr
Arm/Group | NewGam
Number analyzed (Participants) | 51
Serious infections per person-year of tr | 0.080

2. Secondary Outcome: IgG Trough Level Concentration
Description: Total IgG trough concentrations were measured in serum samples taken before each infusion.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | NewGam
Number analyzed (Participants) | 51
g/L
  Infusion 1 | 9.91 (2.845)
  Termination visit | 10.32 (3.429)

3. Secondary Outcome: Trough Level Concentration of Antibodies Against Haemophilus Influenzae
Description: Trough level concentrations of antibodies against Haemophilus influenzae were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | NewGam
Number analyzed (Participants) | 51
µg/mL
  Infusion 1 | 1.96 (1.473)
  Termination visit | 2.51 (1.765)

4. Secondary Outcome: Trough Level Concentration of Antibodies Against Measles
Description: Trough level concentrations of antibodies against measles were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | NewGam
Number analyzed (Participants) | 51
mIU/mL
  Infusion 1 | 854.08 (455.220)
  Termination visit | 1257.76 (706.276)

5. Secondary Outcome: Trough Level Concentration of Antibodies Against Streptococcus Pneumoniae
Description: Trough level concentrations of antibodies against Streptococcus pneumoniae (serotypes types 6B, 14, 9V, 18C, 19F, 4, and 23F) were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | NewGam
Number analyzed (Participants) | 51
µg/mL
  Infusion 1 - serotype 4 | 1.03 (0.680)
  Termination visit - serotype 4 | 1.10 (0.673)
  Infusion 1 - serotype 6B | 1.97 (1.226)
  Termination visit - serotype 6B | 2.10 (1.134)
  Infusion 1 - serotype 9V | 1.86 (0.938)
  Termination visit - serotype 9V | 1.95 (0.942)
  Infusion 1 - serotype 14 | 7.21 (4.355)
  Termination visit - serotype 14 | 7.97 (5.057)
  Infusion 1 - serotype 18C | 2.28 (2.234)
  Termination visit - serotype 18C | 2.38 (2.077)
  Infusion 1 - serotype 19F | 6.56 (4.272)
  Termination visit - serotype 19F | 6.41 (3.843)
  Infusion 1 - serotype 23F | 1.87 (1.102)
  Termination visit - serotype 23F | 2.03 (0.918)

6. Secondary Outcome: Trough Level Concentration of Antibodies Against Cytomegalovirus
Description: Trough level concentrations of antibodies against cytomegalovirus were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: U
Arm/Group | NewGam
Number analyzed (Participants) | 51
U
  Infusion 1 | 30.75 (6.823)
  Termination visit | 30.16 (6.670)

7. Secondary Outcome: Trough Level Concentration of Antibodies Against Tetanus
Description: Trough level concentrations of antibodies against tetanus were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | NewGam
Number analyzed (Participants) | 51
IU/mL
  Infusion 1 | 2.70 (1.467)
  Termination visit | 2.37 (1.389)

8. Secondary Outcome: Trough Level Concentration of Antibodies Against Varicella-zoster Virus
Description: Trough level concentrations of antibodies against varicella-zoster virus were measured in serum blood samples collected before the 1st infusion in all participants, before the 9th and 10th infusions in participants receiving NewGam every 3 weeks, before the 7th and 8th infusions in participants receiving NewGam every 4 weeks, and at the termination visit for all participants.
Time Frame: Baseline to end of the study (up to 12 months)
Population: Pharmacokinetic set: All participants who had concentration data for at least 1 of the pre-infusion IgG trough levels.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | NewGam
Number analyzed (Participants) | 51
U/mL
  Infusion 1 | 125.13 (36.490)
  Termination visit | 119.02 (40.457)

9. Secondary Outcome: Total Number of Infections
Description: The number of infections included serious bacterial infections (bacterial pneumonia, bacteraemia/sepsis, osteomyelitis/septic arthritis, visceral abscess, bacterial meningitis) and other infections. For other infections, the Medical Dictionary for Regulatory Activities (MedDRA) preferred term was used to determine the type of infection. They were grouped into the following categories as determined by a medical expert: Ear infections, eye infections, infections of the gastrointestinal tract, infections of the genitourinary tract, upper respiratory tract infections, lower respiratory tract infections, infections of the skin, and infections not elsewhere classified.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Infections
Arm/Group | NewGam
Number analyzed (Participants) | 51
Infections | 189

10. Secondary Outcome: Number of Non-serious Infections
Description: The MedDRA preferred term was used to determine the type of non-serious infection. They were grouped into the following categories as determined by a medical expert: Ear infections, eye infections, infections of the gastrointestinal tract, infections of the genitourinary tract, upper respiratory tract infections, lower respiratory tract infections, infections of the skin, and infections not elsewhere classified. The total number of infections and the number in each category are reported.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Infections
Arm/Group | NewGam
Number analyzed (Participants) | 51
Infections
  All infections | 185
  Ear infections | 13
  Eye infections | 4
  Infections of the gastrointestinal tract | 28
  Infections of the genitourinary tract | 14
  Upper respiratory tract infections | 90
  Lower respiratory tract infections | 16
  Infections of the skin | 5
  Infections not elsewhere classified | 14

11. Secondary Outcome: Time to Resolution of Serious and Other Infections
Description: Since infections were reported as adverse events, the time to resolution of an infection was the time from the start date of the infection adverse event to the end date of the infection adverse event.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NewGam
Number analyzed (Participants) | 51
Days
  Serious infections | 14.3 (7.63)
  Other infections | 18.4 (34.82)

12. Secondary Outcome: Percentage of Participants Treated With Antibiotics
Description: The total percentage of participants treated with antibiotics, as well as, the percentage of participants treated with antibiotics therapeutically and prophylactically are reported.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 51
Percentage of participants | 82.4

13. Secondary Outcome: Number of Antibiotic Treatment Episodes Per Person-year of Treatment
Description: The number of antibiotic treatment episodes per person-year of treatment was calculated by the following formula: Total number of antibiotic treatment episodes / patient-years of NewGam treatment.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Treatment episodes/person/year
Arm/Group | NewGam
Number analyzed (Participants) | 51
Treatment episodes/person/year | 3.045

14. Secondary Outcome: Number of Antibiotic Treatment Days Per Person-year of Treatment
Description: The number of antibiotic treatment days per person-year of treatment was calculated by the following formula: Total number of antibiotic treatment days / patient-years of NewGam treatment.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Treatment days/person/year
Arm/Group | NewGam
Number analyzed (Participants) | 51
Treatment days/person/year | 87.301

15. Secondary Outcome: Number of Participants Hospitalized Due to an Infection
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NewGam
Number analyzed (Participants) | 51
Participants | 1

16. Secondary Outcome: Percentage of Participants With at Least 1 Episode of Fever
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 51
Percentage of participants | 21.6

17. Secondary Outcome: Percentage of Participants That Missed School or Work Due to an Infection
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | NewGam
Number analyzed (Participants) | 51
Percentage of participants | 49.0

18. Secondary Outcome: Changes in the Physical and Psychosocial Child Health Questionnaire-Parent Form Scores From Baseline to the End of the Study
Description: The Quality of Life (QoL) questionnaire Child Health Questionnaire-Parent Form (CHQ-PF50) was completed by a parent or guardian in study participants < 14 years of age. The CHQ-PF50 consists of 50 items organized into 15 subscales.The 15 subscales could be combined into 2 summary scores, physical and psychosocial. The calculated summary scores were transformed to a range of 0-100, where a higher score indicates more positive functioning or better health status. A positive change score indicates improvement.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | NewGam
Number analyzed (Participants) | 17
Units on a scale
  Physical | 2.77 (9.89)
  Psychosocial | 0.26 (7.19)

19. Secondary Outcome: Changes in the Physical and Mental Short Form-36 Health Survey Scores From Baseline to the End of the Study
Description: The Quality of Life (QoL) questionnaire Short Form-36 Health Survey (SF-36-HS) was completed by participants ≥ 14 years of age. The SF-36-HS consists of 36 items organized into 8 subscales. The 8 subscales could be combined into 2 summary scores, physical and mental. The calculated summary scores were transformed to a range of 0-100, where a higher score indicates better health. A positive change score indicates improvement.
Time Frame: Baseline to end of the study (up to 12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | NewGam
Number analyzed (Participants) | 30
Units on a scale
  Physical | -2.23 (9.96)
  Mental | 2.59 (9.63)

ADVERSE EVENTS:
Description: Safety analysis set: All participants who received at least part of 1 treatment with NewGam.
Arm/Group | NewGam
Serious Adverse Events (participants affected / at risk) | 5/51
Other Adverse Events (participants affected / at risk) | 45/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NewGam (N=51)
Gout (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Septoplasty (Surgical and medical procedures) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NewGam (N=51)
Conjunctivitis (Eye disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 10
Pain (General disorders) | 3
Pyrexia (General disorders) | 11
Acute sinusitis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 8
Gastroenteritis viral (Infections and infestations) | 3
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 13
Oral herpes (Infections and infestations) | 3
Otitis media (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 6
Pharyngitis streptococcal (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 15
Viral infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 14
Migraine (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.